CLINICAL TRIAL: NCT03676426
Title: Comparison of a Web-based Advance Directive to a Standard Advance Directive: Randomized Evaluation
Brief Title: Comparison of a Web-based Advance Directive to a Standard Advance Directive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 829211
Record Dates: First submitted 2018-09-07; First posted 2018-09-18 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: GI Cancer; Thoracic Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Advance Care Planning; Advance Directives

STUDY DESIGN:
Masking Description: Patients will be blinded to the comparison being made, but not to the intervention in their arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based AD (Experimental): Patients will be encouraged to use the web platform for advance care planning/advance directive to document their care preferences..
  Interventions: Other: Web platform for advance care planning/advance directive
- Paper AD (Active Comparator): Patients will be given the standard advance directive and encouraged to complete on their own.
  Interventions: Other: Standard advance directive

INTERVENTIONS:
Other: Web platform for advance care planning/advance directive — Ourcarewishes (OCW) is a web-based platform to document advance care planning based at Penn. OCW contains more detailed content on preferences and values than a standard advance directive and allows electronic sharing with loved ones and transmission to the Penn EHR.
  Other Names: ourcarewishes.org
  Arms: Web-based AD
Other: Standard advance directive — Patients receive a paper copy of an advance directive used by social workers at Penn Medicine and are encouraged to complete on their own.
  Arms: Paper AD

SUMMARY:
This study will compare a web-based advance directive to a standard advance directive.

DETAILED DESCRIPTION:
Patients with GI and thoracic malignancies will be randomized to either a standard paper advance directive or the web advance directive (Ourcarewishes.org). Patients will be approached in the Cancer Center and provided the AD information to complete on their own. They will complete a survey at enrollment and a follow up survey administered by email. The primary endpoint will be proportion with new documentation in the EHR at 8 weeks. Second endpoints will include the change in satisfaction with end-of-life plans, AD acceptability, self-reported rates of completion, self-reported rate of sharing with their preferred surrogate decision-maker, proportion with new documentation of preferred decision-maker in the chart, and qualitative feedback. Patients in both groups will receive follow up reminder emails encouraging them to complete the advance directive.

ELIGIBILITY:
Inclusion Criteria (any of the following)

* Pancreatic cancer, any stage except stage 0 (C25),
* NSCLC, stage IIIA or higher (C34),
* SCLC, any stage (C34),
* Colon cancer, stage IIIB or greater (C18),
* Rectal cancer, stage IIB or greater (C21),
* Esophageal cancer (adeno or squamous), any stage (C15),
* Stomach cancer, stage IIB or greater (C16),
* Gallbladder cancer, stage I or greater (C23),
* Cholangiocarcinoma, any stage (C22.1),
* HCC, any stage (no plan for transplant) (C22.0),
* Malignant carcinoid of GI tract, stage IV (C7A.019).

Exclusion criteria:

* Does not have an active patient portal (MyPennMedicine) account,
* Does not use email at least once per month,
* Has already completed a living will,
* Does not speak fluent English,
* Unwilling to be contacted by email,
* Determined to be too ill or inappropriate for participation by patient's oncologist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
New documentation of advance care planning in the EHR | 8 weeks
  any new advance directive or advance care planning note, excluding an advance directive that either 1) contains only information on the patient's preferred surrogate decision-makers, or 2) is blank except for personal identifying information.

SECONDARY OUTCOMES:
Change in satisfaction with end-of-life plans | Initial completed at enrollment, survey sent again at 15 days
  Change in mean score on the satisfaction with end-of-life scale, adapted from doi: 10.1377/hlthaff.2012.0895, Canadian Healthcare Evaluation Project (CANHELP) questionnaire. This scale measures satisfaction with end-of-life planning on a 12-60 point scale (if all questions answered, 0 possible if "don't know/refusal" chosen for all 12 questions. Higher scores are considered better.
Acceptability | Survey sent at 15 days (reminders at 2 week intervals x 2, then phone call)
  Mean score on an acceptability scale adapted from DOI: 10.1016/j.pec.2007.08.015. This is a scale that measures advance directive acceptability on a 5-50 point scale. Higher scores represent better outcomes.
Self reporting sharing with surrogate | Survey sent at 15 days (reminders 4, 6)Survey sent at 15 days (reminders at 2 week intervals x 2, then phone call)
  Proportion reporting sharing with preferred surrogate
Self reporting completion | Survey sent at 15 days (reminders at 2 week intervals x 2, then phone call)
  Proportion reporting completing some or all of the advance directive
Qualitative feedback | Survey sent at 15 days (reminders at 2 week intervals x 2, then phone call)
  Comments on what patients liked, did not like, and would change about the advance directive
Surrogate preferences | 8 weeks
  Proportion of subjects with new information about their preferred surrogate decision-maker in the chart

CONTACTS AND LOCATIONS:
Locations (1):
- Ruth & Raymond Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Halpern SD, Loewenstein G, Volpp KG, Cooney E, Vranas K, Quill CM, McKenzie MS, Harhay MO, Gabler NB, Silva T, Arnold R, Angus DC, Bryce C. Default options in advance directives influence how patients set goals for end-of-life care. Health Aff (Millwood). 2013 Feb;32(2):408-17. doi: 10.1377/hlthaff.2012.0895. PMID 23381535
- [Background] Sudore RL, Landefeld CS, Barnes DE, Lindquist K, Williams BA, Brody R, Schillinger D. An advance directive redesigned to meet the literacy level of most adults: a randomized trial. Patient Educ Couns. 2007 Dec;69(1-3):165-95. doi: 10.1016/j.pec.2007.08.015. Epub 2007 Oct 17. PMID 17942272